CLINICAL TRIAL: NCT07121816
Title: Use of the ECG Watch in Palpitation Assessment: Feasibility Study
Acronym: WATCH-RHYTHM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hôpital Haut-Lévêque (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2023 ABU ALRUB
Record Dates: First submitted 2025-06-26; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Palpitation
Keywords: Palpitations; ScanWatch (Withings®); ECG

STUDY DESIGN:
Intervention Model Description: ScanWatch (Withings®) For a minimum of 14 days to 1 month, the patient will wear the connected watch, and activate it during an attack of palpitations. For 14 days, he will be concomitantly equipped with a Spider Flash.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using a 24-hour Holter ECG and a smartwatch (Experimental): A single group of patients, all using a 24-hour Holter ECG and a smartwatch
  Interventions: Device: ECG watch

INTERVENTIONS:
Device: ECG watch — ECG watch in palpitation assessment

SUMMARY:
Palpitations are the cause of 16% of reasons for consultation with the general practitioner. 41% of palpitations are secondary to cardiac arrhythmia. If a rhythm or conduction disorder is recorded in a symptomatic context, then the cardiac origin can be validated or invalidated. The challenge therefore consists of obtaining an ECG trace during an attack of palpitations (per-critical ECG). Since patients are rarely symptomatic during consultations, additional exploration by ambulatory electrocardiographic recording is essential. To date, the 24-hour Holter ECG is currently the most used in current practice, only has a sensitivity of 22 to 35% maximum depending on the studies. We hypothesize that the ECG watch is a reliable medical tool in the etiological assessment of palpitations, with at least 90% of traces interpretable.

The main objective of this study is to validate the use of the ScanWatch watch (Withings®) in the assessment of palpitations.

DETAILED DESCRIPTION:
The following examinations will be carried out:

* After inclusion: Information on the operation of the connected watch, loan of the watch, and implementation of a 14-day Spider Flash.
* For a minimum of 14 days to 1 month, the patient will wear the connected watch, and activate it during an attack of palpitations. For 14 days, he will be concomitantly equipped with a Spider Flash.
* All of the watch's traces will be automatically transferred to the Withings RPM data visualization platform independent of each center. The traces will then be centralized anonymously to analyze the results.
* At the end of the loan period, the patient then returns the watch to the cardiology department of their reference center. The Spider Flash is removed after 14 days.
* The patient will be summoned to carry out additional examinations or make therapeutic modifications according to the results of these examinations as part of routine care by their reference center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, referred for cardiological consultation for assessment of palpitations, after which an outpatient electrocardiographic exploration is carried out by the cardiologist.
* - Patient presenting at least 1 palpitation attack per month over the last 3 months or at least 1 palpitation attack per week over the last month.
* Patient equipped with a smartphone compatible with the HealthMate application.
* Able to give consent to participate in research.
* Affiliation to a social security regime.

Exclusion criteria :

* Patient physically or mentally unable to make a recording using the connected watch.
* Patient contraindicated for the application of skin patches.
* Patient with pacemaker or defibrillator.
* Pregnant or breastfeeding women
* Patients of legal age under protective supervision
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Concordance between the number of per-critical tracings obtained via the connected watch (explanatory variable) and the number of interpretable tracings obtained (dependent variable) | One month

SECONDARY OUTCOMES:
Average number of traces per critical necessary to obtain an interpretable trace with the Spider Flash and the connected watch. | One month
Average time to obtain a per critical trace | One month
Classification of recorded events | One month
  Device events Cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Saer ABU ALRUB, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France